CLINICAL TRIAL: NCT01900418
Title: Physical Activity to Reduce Joint Pain During Aromatase Inhibitor Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Leigh F Callahan, PhD, Mary Link Briggs Distinguished Professor of Medicine, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 13-2321
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Joint Pain; Breast Cancer
Keywords: breast cancer; aromatase inhibitors; physical activity; joint pain
MeSH Terms: conditions — Arthralgia; Breast Neoplasms; Motor Activity | interventions — Walking; methyl hydroxyethyl cellulose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Walking (Active Comparator): Walk with Ease
  Interventions: Behavioral: Walk with Ease
- Wait list control (No Intervention): Wait list control receiving the active intervention 6 weeks later.

INTERVENTIONS:
Behavioral: Walk with Ease — An evidence-based walking program
  Arms: Walking

SUMMARY:
For post-menopausal women diagnosed with hormone-receptor positive breast cancer tumors, aromatase inhibitors (AIs) are the standard adjuvant hormone treatment to prolong disease-free survival and time-to-recurrence. Unfortunately, joint pain/stiffness/achiness (arthralgia) is a common side-effect of AIs. This "proof-of-concept" study explores how an evidence-based physical activity (PA) program- the Arthritis Foundation's Walk with Ease (WWE) program- can be adapted for breast cancer survivors on AI therapy to: 1) Help them maintain or achieve recommended levels of PA, 2) reduce their joint pain/stiffness/achiness, and 3) thereby enable them to remain on AI therapy as prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Taking an aromatase inhibitor as adjuvant treatment for State I, II, or II breast cancer for at least 4 weeks
* Experiencing more than mild joint pain/symptoms
* 21 or older
* have permission from physician to engage in moderate intensity physical activity

Exclusion Criteria:

* Undergoing chemotherapy and/or radiation therapy at any time during the study period
* Scheduled for major surgery during the study period
* Presently engaged in high levels of physical activity on a daily basis
* Less than 21 years of age
* Unable to walk or engage in moderate intensity physical activity

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Self-reported joint pain | 6 weeks
  A valid and reliable 10cm Visual Analog Scale will be used to assess self-reported joint pain. This scale has been used in numerous trials.

SECONDARY OUTCOMES:
Self-reported walking | 6 weeks
  This will be measured by the number of days walked per week and the number of minutes per walk.

OTHER OUTCOMES:
Self-reported fatigue | 6 weeks
  A valid and reliable Visual Analog Scale will be used to assess fatigue.
Self-reported joint stiffness | 6 week
  A valid and reliable Visual Analog Scale will be used to assess joint stiffness.
Pain | 6 weeks
  The Brief Pain Inventory Short Form will be used to assess pain. It is a valid and reliable instrument that has been used in other studies of breast cancer survivors.
Lower extremity pain and function | 6 weeks
  The Western Ontario McMaster Universities Arthritis Index will be used to assess hip and knee pain and function.
Quality of life | 6 weeks
  Functional Assessment of Cancer Therapy-General (FACT-G)
Beliefs about engaging in exercise | 6 weeks
  Expectations for Exercise (OEE) scale
Self-efficacy to manage joint pain | 6 weeks
  Arthritis Self-Efficacy Scale (ASE)
Engagement in Physical Activity | 6 weeks
  Behavioral Risk Factor Surveillance System (BRFSS) Questionnaire 2011
Helplessness | 6 weeks
  Rheumatology Attitudes Index (RAI)
Adverse event | 6 weeks
  Self-report of any adverse events will be used to monitor safety.
Feasibility | 6 weeks
  Achievement of 100% recruitment of the enrollment target and 80% completion will indicate program feasibility.
Tolerability | 6 weeks
  Self-report of engaging in any walking level during the 6 week period by 50% of participants will indicate tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh F Callahan, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States